CLINICAL TRIAL: NCT06992830
Title: Cardioneuroablation of Atrial Ganglionated Plexi in Patients With Variant Angina
Brief Title: Cardioneuroablation for Variant Angina
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhibing Lu (Other)
Responsible Party: Sponsor-Investigator, Zhibing Lu, The chief of cardiology department, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025032
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-05

CONDITIONS: Variant Angina
MeSH Terms: conditions — Angina Pectoris, Variant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardioneuroablation group (Experimental): Participants diagnosed with medication-refractory variant angina or those unable or unwilling to take medications regularly will undergo a catheter-based cardioneuroablation (CNA) procedure. CNA targets epicardial cardiac ganglionated plexi (GP), which are clusters of autonomic ganglia involved in parasympathetic modulation of cardiac function. The procedure is designed to reduce parasympathetic overactivity contributing to coronary artery spasms. Ablation will be performed using a radiofrequency catheter to eliminate GP areas identified by anatomical landmarks and electrophysiological mapping. No control or sham procedure is included in this single-arm study.
  Interventions: Procedure: cardioneuroablation

INTERVENTIONS:
Procedure: cardioneuroablation — Participants diagnosed with medication-refractory variant angina or those unable or unwilling to take medications regularly will undergo a catheter-based cardioneuroablation (CNA) procedure. CNA targets epicardial cardiac ganglionated plexi (GP), which are clusters of autonomic ganglia involved in parasympathetic modulation of cardiac function. The procedure is designed to reduce parasympathetic overactivity contributing to coronary artery spasms. Ablation will be performed using a radiofrequency catheter to eliminate GP areas identified by anatomical landmarks and electrophysiological mapping. No control or sham procedure is included in this single-arm study.

SUMMARY:
Variant angina, also known as vasospastic angina, is a form of chest pain caused by temporary spasms of the coronary arteries, which reduce blood flow to the heart. These spasms often occur at rest and may lead to serious complications, including life-threatening heart rhythm problems and sudden cardiac death. While most patients improve with medications such as calcium channel blockers and nitrates, some continue to have symptoms despite treatment. In addition, some patients are unable or unwilling to take medications regularly, which further limits effective management. These cases are referred to as medication-refractory or drug-intolerant variant angina.

The autonomic nervous system, which controls involuntary functions like heart rate and blood vessel tone, is believed to play an important role in the development of coronary artery spasms. Recent research suggests that imbalances in autonomic activity, particularly excessive parasympathetic signals, may trigger these spasms.

Cardioneuroablation (CNA) is a minimally invasive procedure that uses a catheter to target specific nerve clusters called cardiac ganglionated plexi, located on the surface of the heart. These plexi are important centers of autonomic control and are mostly made up of parasympathetic nerve cells. Originally developed to treat conditions such as fainting spells and certain types of abnormal heart rhythms, CNA works by selectively reducing abnormal parasympathetic activity in the heart.

This study is designed to explore whether CNA can help relieve chest pain and reduce coronary spasms in patients with variant angina who do not respond to medications or cannot take them consistently. The study will evaluate the safety, practicality, and potential benefits of this approach as a new treatment option for a difficult-to-manage heart condition.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years;
* variant angina;
* positive ergonovine provocation test;
* refractory to antispasmodic drug therapy, or inability to achieve adequate symptom control due to drug intolerance, poor adherence, or unwillingness to take medications regularly.

Exclusion Criteria:

* cardiogenic shock;
* chronic heart failure;
* life expectancy less than 12 months;
* current participation in another clinical study without completing the primary endpoint visit; inability to provide informed consent;
* women of childbearing potential without effective contraception or who are breastfeeding;
* coronary artery stenosis ≥50% or FFR ≤0.80;
* sick sinus syndrome or high-degree AV block without pacemaker;
* systolic blood pressure <90mmHg or heart rate <50 bpm;
* allergy to diltiazem, nitrates, or nitroglycerin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency of Coronary Spasm Episodes | Baseline and up to 6 months post-procedure
  The number of coronary spasm episodes will be recorded before and after the procedure using 24-hour Holter ECG and integrated dynamic ECG device. Reduction in episode frequency will be used to evaluate treatment efficacy.
Change in Angina Attack Frequency | Baseline and up to 6 months after treatment
  The frequency of chest pain episodes will be assessed through patient diaries and clinical interviews to evaluate symptom relief after treatment.
Severity of Coronary Spasms | Baseline and up to 6 months post-procedure
  Severity will be assessed using imaging findings and clinical scoring systems, such as the Canadian Cardiovascular Society (CCS) Angina Grading Scale, to compare pre- and post-procedural status. CCS Angina Grading Scale ranges from Class I (least severe) to Class IV (most severe), with higher scores indicating worse angina severity. Additional imaging-based assessments (e.g., degree of coronary artery narrowing on angiography) will be qualitatively or semi-quantitatively described.
Electrocardiographic Changes | Baseline and up to 6 months
  Standard 12-lead ECGs and 24-hour Holter monitoring will be analyzed for changes in ST-segment shifts and arrhythmias before and after the procedure.
Major Adverse Cardiovascular Events | From procedure until 6 months post-procedure
  Incidence of cardiovascular events including arrhythmia, cardiac arrest, cardiac death, and acute myocardial infarction will be recorded during follow-up.
Heart Rate Variability (HRV) Changes | Baseline and 1, 3, and 6 months post-treatment
  HRV parameters will be analyzed from 24-hour Holter ECG to assess autonomic modulation following ablation.
Requirement for Anti-Anginal Medications | Baseline and up to 6 months post-procedure
  Dosage and frequency of anti-anginal drug use will be recorded to assess dependence on medication after CNA.

SECONDARY OUTCOMES:
Acute Procedural Success Rate | Intraoperative (immediate post-procedure)
  Defined as successful identification and ablation of ganglionated plexi without intraoperative complications.
Incidence of Acute Procedural Complications | Within 24 hours post-procedure
  Includes intraoperative events such as vascular injury, pericardial effusion, and procedural arrhythmias.
Short-term Postoperative Complications | Up to 30 days post-procedure
  Includes post-procedural complications such as bleeding, infection, and arrhythmias.
Mid- to Long-Term Complications | From 30 days to 12 months post-procedure
  Includes recurrence of coronary spasm, new myocardial infarction, and worsening of cardiac function.
Biomarker Monitoring (e.g., Cardiac Enzymes and Inflammatory Markers) | Baseline and within 72 hours post-procedure
  Serum levels of specific biomarkers will be measured to evaluate myocardial injury and systemic inflammation. These include cardiac enzymes (e.g., troponin I/T, CK-MB) and inflammatory markers (e.g., C-reactive protein [CRP], interleukin-6 [IL-6]). Blood samples will be collected at baseline and within 72 hours post-ablation. Levels will be quantified using standard laboratory assays, and changes will be compared to evaluate procedure-related biological responses.
Comparison of parameters related to coronary vasospasm induced by ergonovine provocation testing before and after CNA | Periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China